CLINICAL TRIAL: NCT05774548
Title: Epidemiological Impact and Cost-effectiveness of Long-acting Antiretrovirals for Pre-exposure Prophylaxis Among Key Populations in Thailand
Brief Title: LA PrEP Impact and Cost-effectiveness (TEAMS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of HIV Research and Innovation Foundation, Thailand (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IHRI019
Record Dates: First submitted 2023-02-22; First posted 2023-03-17 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Hiv
Keywords: HIV, PrEP
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- (PHASE I) Attributes identification (Experimental): To identify attributes of importance for our research question and assign possible levels to these attributes, a combination of literature review and qualitative approaches will be conducted
  Interventions: Other: In-depth interviews (IDI); Other: Focus group discussion (FGD)

INTERVENTIONS:
Other: In-depth interviews (IDI) — In-depth interviews (IDI) 20 MSM,20 TGW, current, previous PrEP users will assess which attributes are relevant each population. Posters will be used to recruit for IDIs. Self-reported HIV-negative who either report interest in current or past PrEP use will be eligible to participate in IDI. IDI will be conducted by a study by in-person, on-line interviews.
Other: Focus group discussion (FGD) — Focus group discussion (FGD) will discuss a interested information from IDIs. IDIs will be informed, invited to a FGD. FGD recruit 6-10 IDI. 10 random number will be generated using statistical if more 10 individuals show interest in participating in a FGD. If there are less than 6 accepted participants for a FGD, the backup list or new participant will be invited. Study will perform FGD by in-person, on-line conference. Data obtained during a process will be used to create a list of attributes for each population, their levels to include in the choice tasks, ensuring that a choices are plausible, exchangeable.

SUMMARY:
This study will have three components:

1. Discrete choice experiments
2. Analysis of routine service data
3. Impact and cost-effectiveness analyses using results from 1 and 2

DETAILED DESCRIPTION:
Discrete choice experiments (DCE) will be part of a survey, assessing sociodemographic characteristics, risk behavior, PrEP related information. Two separate surveys and DCEs will be designed, one for MSM, and one for TGW. Information collected through DCEs will allow us to estimate user values in the absence of observations or readily available data, and use these preferences to inform mathematical modeling on the impact and cost-effectiveness of long-acting PrEP. DCEs will be designed as per best-practice guidance by the International Society for Pharmacoeconomics and Outcomes Research (ISPOR). To maximize statistical and response efficiency, the number of attributes selected for evaluation must be restricted, i.e. the most important attributes must be known prior to construction. Therefore, the DCE design and implementation of the survey will be conducted in different phases:

PHASE I - Identification of attributes In-depth interviews (IDIs) with up to 40 potential, current, previous PrEP users (20 MSM,20 TGW) will assess which attributes are most relevant among each population. Posters will be used to recruit participants for IDIs. Self-reported HIV-negative MSM, TGW who either report interest in PrEP use, current PrEP use, or past PrEP use, will be eligible to participate in the IDIs. IDIs will be conducted by the study staff by in-person or on-line interviews. Focus group discussion (FGD) will prepare to discuss the interested information from IDIs. Following IDIs, participants will be informed and invited to the focus group discussion. A FGD will recruit 6-10 IDI participants from each MSM, TGW group. A list of 10 random numbers will be generated using statistical software if more than 10 individuals show interest in participating in the FGD. If there are less than 6 accepted participants for the FGD, the backup list or a new participant will be invited. The study staff will perform FGD by in-person or on-line conference. Data obtained during this process will be used to create a final list of attributes for each population and their levels to include in the choice tasks, ensuring that the choices are plausible and exchangeable. The number of DCE choice sets will be about 6 per person.

PHASE II - Pilot testing of DCE (The result from Phase I will be used for finalize an initial draft in this part) Initial drafts of the choice tasks (one draft for MSM and one draft for TGW) will be administered to convenience samples of 30 MSM, 30 TGW (10% of phase III sample size), respectively, to obtain feedback about difficulty of tasks, plausibility of levels, length, wording and clarity using a survey form. Final DCEs for each population will be agreed upon by consensus, and incorporated in the surveys.

PHASE III - Survey implementation (The result from Phase II will be used for finalize a survey in this part).

Two final surveys will be launched:1 survey for MSM, 1 survey for TGW. Both surveys will collect data on:

1. Participant information, including:

   1. Sociodemographic information
   2. Risk behavior
   3. HIV testing
   4. STI testing and diagnoses
2. PrEP knowledge and use

   1. Awareness of different PrEP modalities
   2. Interest in different PrEP modalities
   3. Preferences for different PrEP modalities
   4. Current and past use
3. DCE of different PrEP options. Although the final list of attributes will be based on literature review and interviews, potential attributes of interest and their levels are:

   1. Product form (oral, injectable)
   2. Dosing frequency (daily, once every 2 months, once every 6 months, once every 12 months)
   3. Type of facility (hospital, CBO, primary care center, pharmacy, home)
   4. Type of provider preference (KP lay provider, doctor, nurse, pharmacist, self)
   5. Monthly cost out of pocket (free, up to 500 THB, up to 1000 THB)
   6. Side effects (mild, moderate)

Data from these surveys will be analyzed to identify the most important drivers for PrEP preference. This will allow us to analyze the trade-offs that respondents make, to quantitatively explore what drives individual decision making and the relative strength of preferences. These findings will be used to project the hypothetical uptake of long acting antiretrovirals with different characteristics, the impact of this formulation on the uptake of oral PrEP, and how certain long acting antiretroviral characteristics will affect the uptake. Findings generated will be used to conduct epidemiological impact and cost-effectiveness analyses. Uptake projections will be determined for those never using PrEP before, for those having used oral PrEP before and stopped, and for those currently using oral PrEP.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years
* Individual assigned male at birth reporting sex with men in the past 12 months
* Self-reported HIV-negative MSM and TGW who either report interest in PrEP use, current PrEP use, or past PrEP use
* Permit audio recording during the interview and/or discussion.

Exclusion Criteria:

* Not willing to participate in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10720 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The epidemiological impact of long-acting antiretrovirals for HIV prevention among Thai MSM and TGW at risk of HIV infection | 12 months
  Epidemiological impact analyses will compare a current scenario in which PrEP is only available as an oral formulation to a scenario in which long-acting PrEP is also available.
The cost-effectiveness of long-acting antiretrovirals for HIV prevention among Thai MSM and TGW at risk of HIV infection | 12 months
  The cost-effectiveness analysis will be based on previous HIV transmission models published by the Erasmus Medical Centre

SECONDARY OUTCOMES:
Proportion of MSM and TGW indicating uptake of PrEP in hypothetic scenarios, impact of sociodemographic and behavioral characteristics on projected uptake | 18 months
  The uptake of different PrEP modalities will be measured via a discrete choice experiment survey with clients in KP-led PrEP clinic
Preferred PrEP modalities among Thai MSM and TGW, trade-off of different PrEP attributes | 18 months
  To quantify preference for long-acting antiretrovirals as PrEP in Thai MSM and TGW using discrete choice experiments
Patterns of PrEP use | 18 months
  Patterns of PrEP use will analyze from the data such as discontinuation rates and restarts of oral PrEP in KP-led PrEP program

CONTACTS AND LOCATIONS:
Overall Officials: Nittaya Phanuphak, MD,PhD., Principal Investigator — INSTITUTE OF HIV RESEARCH AND INNOVATION FOUNDATION
Locations (12):
- Thailand (12):
  - Rainbow Sky Association of Thailand (RSAT), Bangkok, Bangkapi
  - The Service Workers In Group Foundation (SWING), Bangkok, Building 3, Patpong, Surawong Road
  - The Service Workers In Group Foundation (SWING), Bang Lamung, Changwat Chon Buri
  - Rainbow Sky Association of Thailand (RSAT), Chon Buri, Changwat Chon Buri
  - Rainbow Sky Association of Thailand (RSAT), Hat Yai, Changwat Songkhla
  - Tangerine Clinic, Bangkok, Pathumwan
  - The Service Workers In Group Foundation (SWING), Bangkok, Phay Thai
  - CAREMAT, Chiang Mai
  - Mplus Foundation, Chiang Mai
  - Mplus Foundation, Chiang Rai
  - Mplus Foundation, Phitsanulok
  - Rainbow Sky Association of Thailand (RSAT), Ubon Ratchathani

REFERENCES:
- See also: The epidemiological impact and cost-effectiveness of key population-led PrEP delivery to prevent HIV among men who have sex with men in Thailand: A modelling study — https://doi.org/10.1016/j.lansea.2022.100097